CLINICAL TRIAL: NCT01109498
Title: A Study to Determine the Safety and Efficacy in Lipoprotein Lipase-Deficient Subjects After Intramuscular Administration of AMT-011, an Adeno-Associated Viral Vector Expressing Human Lipoprotein LipaseS447X
Brief Title: Safety and Efficacy in LPL-Deficient Subjects of AMT-011, an Adeno-Associated Viral Vector Expressing Human Lipoprotein Lipase [S447X]
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam Molecular Therapeutics (Industry)
Collaborators: International Antiviral Therapy Evaluation Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-011-01
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2010-04

CONDITIONS: Familial Lipoprotein Lipase Deficiency
Keywords: LPLD; Lipoprotein Lipase Deficiency; Chylomicronaemia; Genetherapy; AAV; Alipogene Tiparvovec; AMT-011; Lipoprotein Lipase
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Alipogene tiparvovec; Mycophenolic Acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose cohort 3 x 10^11gc/kg (Experimental): intra muscular, 3 x E11 gc per kg body weight, injected in a single series of intramuscular injections
  Interventions: Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X]
- Alipogene Tiparvovec, Human LPL [S447X] (Experimental): intra muscular, 3 x E11 gc per kg body weight, injected in a single series of intramuscular injections with immunosuppressants
  Interventions: Drug: Mycophenolate mofetil; Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X]; Drug: cyclosporine
- Alipogene Tiparvovec, Human LPL [S447X], 1xE12 gc/kg (Experimental): intra muscular, 1 x E12 gc per kg body weight, injected in a single series of intramuscular injections with immunosuppressants
  Interventions: Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X]

INTERVENTIONS:
Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X] — intra muscular, 1 x E12 gc per kg body weight, injected in a single series of intramuscular injections
  Other Names: Glybera, AMT-011
  Arms: Alipogene Tiparvovec, Human LPL [S447X], 1xE12 gc/kg
Drug: Mycophenolate mofetil — oral, 2 g/day, day -3 till week 12
  Other Names: CellCept
  Arms: Alipogene Tiparvovec, Human LPL [S447X]
Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X] — intra muscular, 3 x E11 gc per kg body weight, injected in a single series of intramuscular injections
  Other Names: Glybera, AMT 011
  Arms: Alipogene Tiparvovec, Human LPL [S447X]; Dose cohort 3 x 10^11gc/kg
Drug: cyclosporine — oral, 3 mg/kg/day, day -3 till week 12
  Other Names: Neoral
  Arms: Alipogene Tiparvovec, Human LPL [S447X]

SUMMARY:
LPLD is a rare autosomal recessive disorder, characterized by the presence of marked chylomicronemia and hence hypertriglyceridemia. Clinically the most severe manifestation of chylomicronemia, is acute pancreatitis, which can be lethal. There is no effective therapy available to modulate the course of the illness and prevent complications for these patients. The current clinical management consists of severe reduction of dietary fat that is hard if not almost impossible to comply with. LPLD subjects continue to experience pancreatitis attacks, and are admitted to intensive care units on several occasions.

Alipogene tiparvovec corrects or restores lipoprotein lipase (LPL) function long term, and hence reverses some symptoms, halts the disease progression and prevents further complications. Alipogene tiparvovec gene therapy ensures that a catabolically beneficial variant of the human LPL gene, LPL[S447X] is expressed and active in the relevant tissues in humans. Delivery of the gene is realized via intramuscular injection of an adeno-associated viral vector, pseudotyped with AAV1 capsids.

DETAILED DESCRIPTION:
The CT-AMT-011-01 study is an open-label, dose-escalating study evaluating the safety and efficacy of a single intramuscular administration of AMT-011 (at multiple sites). The study will be performed in the Community Genomic medicineCenter (CGMC) Chicoutimi, Canada, under the supervision of their medical ethical committee and according to the local biosafety procedures. The study participants will be treated under the responsibility of a Principal Investigator specialised in the treatment of lipid disorders. A total number of 14 subjects will be administered. Participants will be screened 3 weeks prior to administration of AMT-011 and will be evaluated for 12 weeks post administration in this study. After the study, subjects will be followed up long term with particular emphasis on the safety and efficacy aspects of LPL gene therapy using AMT-011. Subjects will be evaluated at the clinical site at 19 weeks, 26 weeks, 39 weeks, 1 year, 1.5 years, 2 years, 3 years, 4 years and 5 years after administration of AMT-011. The TG values that are obtained at week 26 will be used for secondary efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible Population Study participants must have participated in the preceding observation study (Prep-02: Appendix III) and be diagnosed with lipoprotein lipase deficiency, meeting the following criteria: (I) Their lipoprotein lipase activity levels in post-heparin plasma should be ≤20 % of normal; (II) Confirmed homozygocity or compound heterozygocity for mutations in the LPL gene; (III) Post-heparin plasma LPL mass should be >5% of normal; (IV) Median fasting plasma TG concentrations >10.00mmol/L, as determined on the basis of 5 consecutive time points in the preceding observation study with a history of pancreatitis.
* General Health The participant must be in good general physical health with, in the opinion of the investigator, no other clinically significant and relevant abnormalities of medical history, and no abnormalities at the physical examination and routine laboratory evaluation performed prior to the trial.
* Age Age ≥18 years old.
* Sex Male or female. Females must be of non-child bearing potential or with a negative pregnancy test and not breast feeding. Female subjects must use appropriate contraception (if relevant) and their spouse must use barrier contraception for the duration of the study (12 weeks). Males must practice barrier birth control and their spouse should use appropriate contraception until three consecutive semen samples, taken at least 75 days after administration, are negative for AMT-011 vector DNA.
* Compliance The participant is willing to fully comply with all study procedures and requirements of the trial such as restrictions to a low-fat diet (see section 8.1).
* Consent The participant has the mental ability to give voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Disease
* Apolipoprotein CII deficiency.
* Inflammatory muscle disease (e.g. myositis, myopathies or rhabdomolysis).
* Any current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may make the participant unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures (e.g. malignant neoplasia).
* Active infectious disease of any nature, including clinically active viral infections.
* Laboratory Parameters

The following blood screening tests will result in exclusion from participation:

* Platelet count < 100 x 109 /L.
* Hemoglobin < 7.0 mmol/L.
* Liver function disturbances (bilirubin >2.50 x normal, transaminases >3 x ULN).
* CPK > 3 x ULN.
* Creatinine > 3 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of fasting triglyceride (TG) concentrations | 12 weeks
  To achieve a reduction in fasting plasma TG such that the difference in median plasma TG observed before administration and up to 12 weeks after administration represents approximately 40% reduction, on top of a low-fat diet.
safety profile of AMT-011 | 15 years
  Between 6 and 15 years after administration of AMT-011, patients will be annually contacted by phone to monitor delayed adverse events related to administration of AMT-011.

SECONDARY OUTCOMES:
Reduction of TG concentrations | 26 weeks
  To achieve sustained efficacy, defined as approximately 40% reduction in fasting plasma TG up to 26 weeks after administration, on top of a low-fat diet.
Reduction of TG concentrations | 12 weeks
  To achieve a reduction in fasting plasma TG to a level equal to or less than 10.00 mmol/L on top of a low-fat diet at 12 weeks after administration.
Reduction of TG concentrations | 26 weeks
  To achieve sustained efficacy, defined as a reduction in fasting plasma TG at 26 weeks after administration to a level equal to or less than 10.00 mmol/L on top of a low-fat diet.
Biological activity and expression of the transgene product. | 1 year
  To determine the biological activity and expression of the lipoprotein lipase (LPLS447X) transgene product.
Evaluation immune respons | 5 years
  To evaluate potential immune responses against the lipoprotein lipase (LPLS447X) transgene product and the adeno-associated viral (AAV) vector.
To assess the shedding of the viral vector | 1 year
  To assess shedding of AMT-011

CONTACTS AND LOCATIONS:
Locations (1):
- Ecogene-21 Clinical Trial Center/ Centre de santé et de services sociaux de Chicoutimi, Chicoutimi, Quebec, Canada

REFERENCES:
- [Background] Rip J, Nierman MC, Sierts JA, Petersen W, Van den Oever K, Van Raalte D, Ross CJ, Hayden MR, Bakker AC, Dijkhuizen P, Hermens WT, Twisk J, Stroes E, Kastelein JJ, Kuivenhoven JA, Meulenberg JM. Gene therapy for lipoprotein lipase deficiency: working toward clinical application. Hum Gene Ther. 2005 Nov;16(11):1276-86. doi: 10.1089/hum.2005.16.1276. PMID 16259561
- [Background] Ross CJ, Twisk J, Meulenberg JM, Liu G, van den Oever K, Moraal E, Hermens WT, Rip J, Kastelein JJ, Kuivenhoven JA, Hayden MR. Long-term correction of murine lipoprotein lipase deficiency with AAV1-mediated gene transfer of the naturally occurring LPL(S447X) beneficial mutation. Hum Gene Ther. 2004 Sep;15(9):906-19. doi: 10.1089/hum.2004.15.906. PMID 15353045
- [Background] Ross CJ, Liu G, Kuivenhoven JA, Twisk J, Rip J, van Dop W, Excoffon KJ, Lewis SM, Kastelein JJ, Hayden MR. Complete rescue of lipoprotein lipase-deficient mice by somatic gene transfer of the naturally occurring LPLS447X beneficial mutation. Arterioscler Thromb Vasc Biol. 2005 Oct;25(10):2143-50. doi: 10.1161/01.ATV.0000176971.27302.b0. Epub 2005 Jul 7. PMID 16002740
- [Background] Ross CJ, Twisk J, Bakker AC, Miao F, Verbart D, Rip J, Godbey T, Dijkhuizen P, Hermens WT, Kastelein JJ, Kuivenhoven JA, Meulenberg JM, Hayden MR. Correction of feline lipoprotein lipase deficiency with adeno-associated virus serotype 1-mediated gene transfer of the lipoprotein lipase S447X beneficial mutation. Hum Gene Ther. 2006 May;17(5):487-99. doi: 10.1089/hum.2006.17.487. PMID 16716106
- [Background] Stroes ES, Nierman MC, Meulenberg JJ, Franssen R, Twisk J, Henny CP, Maas MM, Zwinderman AH, Ross C, Aronica E, High KA, Levi MM, Hayden MR, Kastelein JJ, Kuivenhoven JA. Intramuscular administration of AAV1-lipoprotein lipase S447X lowers triglycerides in lipoprotein lipase-deficient patients. Arterioscler Thromb Vasc Biol. 2008 Dec;28(12):2303-4. doi: 10.1161/ATVBAHA.108.175620. Epub 2008 Sep 18. No abstract available. PMID 18802015
- [Background] Burnett JR, Hooper AJ. Alipogene tiparvovec, an adeno-associated virus encoding the Ser(447)X variant of the human lipoprotein lipase gene for the treatment of patients with lipoprotein lipase deficiency. Curr Opin Mol Ther. 2009 Dec;11(6):681-91. PMID 20072945
- [Derived] Gaudet D, Methot J, Dery S, Brisson D, Essiembre C, Tremblay G, Tremblay K, de Wal J, Twisk J, van den Bulk N, Sier-Ferreira V, van Deventer S. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: an open-label trial. Gene Ther. 2013 Apr;20(4):361-9. doi: 10.1038/gt.2012.43. Epub 2012 Jun 21. PMID 22717743